CLINICAL TRIAL: NCT01793675
Title: Haplo-identical/Mismatched Hematopoietic Stem Cell Transplantation for Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, Prof., Peking University People's Hospital
Other Study IDs: PUPH IRB [2013] (04)
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Advanced MDS Without Identical Sibling Donor
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- haploidentical transplant: transplant with haploidentical donor
  Interventions: Procedure: transplant with haploidentical donor

INTERVENTIONS:
Procedure: transplant with haploidentical donor — patients with advanced MDS without identical sibling donor receive haploidentical transplant
  Other Names: haploidentical transplant

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) is currently the only curative treatment for myelodysplastic syndrome (MDS), especially for advanced MDS (blast >5%). However, many patients cannot find an HLA-matched donor. haploidentical donor is an alternative stem cell source.

the study hypothesis: Haploidentical/mismatched hematopoietic stem cell transplantation can improve the survival of patients with myelodysplastic syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients with MDS (1)intermediate-2 or high risk (2)low or intermediate-1 risk with drug resistance or disease progression
* without identical sibling donor

Exclusion Criteria:

* Contraindication to HSCT
* Pregnancy
* Mental illness

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with MDS:1)intermediate-2 or high risk 2)low or intermediate-1 risk, drug resistance or disease progression
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2003-04; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
survival rate | participants will be followed for an expected average of one year
  number of participants with survival at one year

SECONDARY OUTCOMES:
incidence of non-relapse mortality | one year
  number of participants with non-relapse mortality at one year

CONTACTS AND LOCATIONS:
Overall Officials: xiaojun huang, M.D., Principal Investigator — Peking University People's Hospital
Locations (8):
- China (8):
  - Nanfang Hospital, Nanfang Medical University, Guangzhou, Guangdong
  - Hebei Tangshan Steel and Iron Company Hospital, Tangshan, Hebei
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - Suzhou University The 1st Affiliated Hospital, Suzhou, Jiangsu
  - Chongqing Medical University The 1st Affiliated Hospital, Chongqing, Sichuan
  - The 3rd Army Medical University The 2nd Affiliated Hospital, Chongqing, Sichuan
  - Peking University People's Hospital, Beijing
  - Aerospace center hospital, Beijing